CLINICAL TRIAL: NCT01102738
Title: The Microbiota of the Premature Neonatal Gastrointestinal Tract: Its Development and Relation to Necrotizing Enterocolitis and Bloodstream Infection
Brief Title: Defining the Intestinal Microbiota in Premature Neonates
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: The Winnicott Foundation (Other); National Heart and Lung Institute (Other); Chelsea and Westminster NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CR01542
Record Dates: First submitted 2010-03-31; First posted 2010-04-13 (Estimated); Results first posted 2020-05-01 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Premature Intestinal Microbiota; Necrotizing Enterocolitis; Late Onset Bloodstream Infection
Keywords: Premature intestinal microbiota; Necrotizing Enterocolitis
MeSH Terms: conditions — Enterocolitis, Necrotizing

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Faecal samples, surplus gut tissue samples (if patient requires bowel resection due to Necrotizing Enterocolitis).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Premature babies (<32 weeks): All premature babies born at less than 32 completed weeks gestation who are admitted to an Imperial College NHS Healthcare Trust Neonatal Intensive Care Unit (St. Mary's Hospital or Queen Charlotte's & Chelsea Hospital), and whose parents/guardians have given their consent will be eligible to enter the study.

SUMMARY:
The investigators will collect daily faecal samples from premature (<32 weeks) infants in the intensive care unit from the day of birth until they are discharged. By using newly developed molecular detection techniques the investigators aim to define more precisely than has ever previously been attempted, all the species of bacteria present in the faeces. This will enable comparison of the pre-morbid and post-morbid intestinal microbiota (all the bacteria in the gut) in premature neonates.

DETAILED DESCRIPTION:
Highly premature infants are susceptible to serious infections such as necrotizing enterocolitis (NEC) and late-onset blood stream infections (BSIs).

NEC is a poorly understood, potentially life-threatening bowel disorder. It is thought that bacteria proliferating abnormally in the bowel may play an important part in its cause, but no single pathogen has yet been identified.

BSIs are commonly caused by gut bacteria. As the highly premature gut is fragile and has increased permeability, poor motility and decreased immune defences, localised inflammation caused by abnormal bacterial growth may allow 'bystander' microbes to translocate through the gut into the blood stream leading to systemic infection.

In a small proportion of infants who develop NEC, surgery will be required as part of treatment of the condition. In these infants the investigators will seek consent to collect a small part of the diseased bowel which has been removed. Similar analysis will be performed on these samples. The analysis of the tissue samples will give us an indication of how well the faeces act as a proxy for the intestinal microbiota.

In this ecological study of the evolution of the intestinal microbiota in preterm infants, by comparing samples from babies who develop NEC or late-onset BSI with those of well babies the investigators will be able to look for differences characteristic of the conditions. This information will help aid design of prevention or treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* All premature babies born at less than 32 completed weeks gestation who are admitted to an Imperial College NHS Healthcare Trust Neonatal Intensive Care Unit (St. Mary's Hospital or Queen Charlotte's & Chelsea Hospital), and whose parents/guardians have given their consent will be eligible to enter the study.

Exclusion Criteria:

* All babies born at more than 32 completed weeks gestation will be excluded from the study.

Max Age: 32 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Premature babies born at less than 32 completed weeks gestation
Sampling Method: Non-Probability Sample
Enrollment: 369 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2013-01 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J Simon Kroll, MA BM FRCP, Principal Investigator — Imperial College London
Locations (3):
- United Kingdom (3):
  - Imperial College London, London
  - Queen Charlotte's and Chelsea Hospital - NICU, London
  - St. Mary's Hospital - Winnicott Baby Unit, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shaw AG, Cornwell E, Sim K, Thrower H, Scott H, Brown JCS, Dixon RA, Kroll JS. Dynamics of toxigenic Clostridium perfringens colonisation in a cohort of prematurely born neonatal infants. BMC Pediatr. 2020 Feb 18;20(1):75. doi: 10.1186/s12887-020-1976-7. PMID 32070310
- [Derived] Sim K, Shaw AG, Randell P, Cox MJ, McClure ZE, Li MS, Haddad M, Langford PR, Cookson WO, Moffatt MF, Kroll JS. Dysbiosis anticipating necrotizing enterocolitis in very premature infants. Clin Infect Dis. 2015 Feb 1;60(3):389-97. doi: 10.1093/cid/ciu822. Epub 2014 Oct 23. PMID 25344536

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Premature Babies (<32 Weeks)
Started | 369
Completed | 369
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Premature Babies (<32 Weeks)
Number analyzed (Participants) | 369
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 369
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: days] | 2 [0 to 14]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 171
  Male | 198
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 339
  Unknown or Not Reported | 28
Region of Enrollment [Number; unit: participants]
  United Kingdom | 369

OUTCOME MEASURES:

1. Primary Outcome: The Composition of Bacteria Present, Established by Ultra-deep RNA Gene Sequencing, in Pre-morbid Faecal Samples From Neonates With Necrotizing Enterocolitis and Late-onset Bacterial Sepsis.
Description: Faecal samples were analysed using 16S rRNA gene sequencing to determine the bacterial content present in faecal samples collected from pre term infants prior to the onset of necrotising enterocolitis.
  Bacteria were identified and relative proportions reported for each faecal sample analysed.
Time Frame: Maximum of 6 months - serial samples collected from each infant (maximum admission duration 6 months), recruitment opened for 24 months.
Population: Faecal samples and clinical data were collected from all participants (369 infants) recruited into the study. Samples were only analysed from infants who developed NEC (n=12) and 3 matched controls (n=36).
Measure: Number; unit: Participants
Arm/Group | Premature Babies (<32 Weeks)
Number analyzed (Participants) | 48
Participants
  Klebsiella OTU associated NEC | 7
  Clostridium associated NEC | 4
  Non Klebsiella or Clostridium associated NEC | 1
  Controls | 36

ADVERSE EVENTS:
Time Frame: Recruitment of infants was over a 24 month period during which adverse event data was collected. All infants were followed up until the end of their admission on the neonatal unit, at which point, data collection ceased. All participants recruited were discharged from the neonatal unit two months from the end of the recruitment period. Time frame over which adverse event data were collected: 26 months
Groups:
- Premature Babies (<32 Weeks): All premature babies born at less than 32 completed weeks gestation who are admitted to an Imperial College NHS Healthcare Trust Neonatal Intensive Care Unit (St. Mary's Hospital or Queen Charlotte's & Chelsea Hospital), and whose parents/guardians have given their consent will be eligible to enter the study.
  No adverse events related to the study occurred. The study was an observational study which only involved the collection of clinical data, faecal samples, urine samples and skin swabs.
Arm/Group | Premature Babies (<32 Weeks)
All-Cause Mortality (participants affected / at risk) | 30/369
Serious Adverse Events (participants affected / at risk) | 0/369
Other Adverse Events (participants affected / at risk) | 0/369

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes